CLINICAL TRIAL: NCT02073344
Title: Prospective Interventional Study Investigating the Effect of Beginning a Renal Replacement Therapy on Obstructive Sleep Apnea and Its Correlation With Overhydration, in End Stage Renal Disease Patients
Brief Title: Effect of Beginning a Renal Replacement Therapy on Obstructive Sleep Apnea in End Stage Renal Disease Patients
Acronym: SASinHD_005
Status: Suspended | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Adam Ogna, Centre d'Investigation et Recherche sur le Sommeil (CIRS), Centre Hospitalier Universitaire Vaudois
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIRS-SASinHD_005
Record Dates: First submitted 2014-02-25; First posted 2014-02-27 (Estimated); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Obstructive Sleep Apnea; End Stage Renal Disease
Keywords: obstructive sleep apnea; overhydration; end stage renal disease; renal transplantation; polysomnography; bioimpedance; leg fluid shift; neck circumference
MeSH Terms: conditions — Sleep Apnea, Obstructive; Kidney Failure, Chronic; Water Intoxication | interventions — Renal Replacement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intevention group (Experimental): A baseline polysomnography (PSG) is performed at inclusion, followed by a follow-up PSG 6 months after the beginning of a renal replacement therapy
  Interventions: Procedure: Renal replacement therapy
- Control group (Experimental): No intervention A baseline polysomnography (PSG) is performed at inclusion, followed by a follow-up PSG at 6 months if the patient is not already on renal replacement therapy
  Interventions: Other: no intervention

INTERVENTIONS:
Procedure: Renal replacement therapy — intermittent hemodialysis or peritoneal dialysis
  Arms: Intevention group
Other: no intervention — no renal replacement therapy
  Arms: Control group

SUMMARY:
The purpose of this study is to investigate the effect of beginning a renal replacement therapy on fluid overload and its consequence on the severity of obstructive sleep apnea, in patients with end stage chronic kidney disease. It aims further to investigate the relationship between overhydration, nocturnal rostral fluid shift and the severity of sleep apnea.

DETAILED DESCRIPTION:
The prevalence of obstructive sleep apnea increases with progressing renal insufficiency. Recent observations suggest a causative relationship between overnight fluid displacement from the legs to the neck soft tissues and the severity of obstructive sleep apnea. We suspect that this pathophysiologic mechanism could explain the increased prevalence of obstructive sleep apnea in patients with fluid overload, including chronic renal failure.

The beginning of a renal replacement therapy modify the fluid balance of the end stage renal disease patients and could therefore impact on the severity of sleep apnea in this population.

The purpose of this trial is to investigate the hypothesis that the transition from untreated end stage renal disease and a renal replacement therapy decreases the severity of sleep apnea, by a reduction of the fluid overload and of the nocturnal rostral fluid shift.

The severity of obstructive sleep apnea is measured by two attended polysomnographies (PSG), a baseline PSG performed before and a follow-up PSG performed 6 month after beginning of a renal replacement therapy. Overhydration and leg fluid are evaluated by bioimpedance, performed at the beginning and at the end of each polysomnography. Patients who have not yet begun a renal replacement therapy 6 months after the baseline PSG will be re-assessed and will be analyzed as control group

ELIGIBILITY:
Inclusion Criteria:

* moderate to severe obstructive sleep apnea, with an apnea-hypopnea index (AHI) ≥ 15/h
* age ≥ 18 years
* patient with end stage renal disease without renal replacement therapy.

Exclusion Criteria:

* unstable congestive heart failure
* active psychiatric disease
* amputation of the lower limbs, proximal to the ankle

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-03; Primary Completion 2021-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
obstructive sleep apnea severity | six months (before and after beginning of a renal replacement therapy)
  Reduction of the obstructive sleep apnea severity, measured by attended polysomnography, six months after beginning of a renal replacement therapy

SECONDARY OUTCOMES:
nocturnal leg fluid volume shift | six months (before and after beginning of a renal replacement therapy)
  Reduction in nocturnal leg fluid volume shift between the legs and the neck, measured by bioimpedance and neck circumference six months after beginning of a renal replacement therapy
relationship between overhydration, leg fluid volume shift, ankle and neck circumference and the severity of obstructive sleep apnea | one night
periodic limb movement disorder (PLMD) | six months (before and after beginning of a renal replacement therapy)
severity of central sleep apnea syndrome | six months (before and after renal beginning of a renal replacement therapy)

CONTACTS AND LOCATIONS:
Overall Officials: Raphaël Heinzer, MD, Principal Investigator — Centre d'Investigation et Recherche sur le Sommeil (CIRS) - Centre Hospitalier Universitaire Vaudois (CHUV); Adam Ogna, MD, Principal Investigator — Centre d'Investigation et Recherche sur le Sommeil (CIRS) - Centre Hospitalier Universitaire Vaudois (CHUV); Valentina Forni Ogna, MD, Principal Investigator — Centre d'Investigation et Recherche sur le Sommeil (CIRS) - Centre Hospitalier Universitaire Vaudois (CHUV)
Locations (1):
- Centre d'Investigation et Recherche sur le Sommeil (CIRS) - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Canton of Vaud, Switzerland